CLINICAL TRIAL: NCT04617067
Title: Phase II, Open Label Clinical Trial of Paricalcitol in Combination With Gemcitabine/ Nab-Paclitaxel Therapy in Advanced Pancreatic Cancer
Brief Title: Paricalcitol Trial: Phase II, Open Label Clinical Trial of Paricalcitol in Combination With Gemcitabine/ Nab-Paclitaxel Therapy in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 19-33; 2020-000073-24 (EudraCT Number); CTRIAL-IE 19-33 (Other: Cancer Trials Ireland ID number)
Record Dates: First submitted 2020-10-27; First posted 2020-11-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced Pancreatic Cancer
MeSH Terms: interventions — paricalcitol; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Patients (Experimental): Open Label: Paricalcitol 12mcg once daily, orally every day of each 28 day cycle PLUS GEM (1000mg/m2) and Nab-paclitaxel (Abraxane®) (125mg/m2) on days 1, 8 and 15 of each cycle.
  Interventions: Drug: Paricalcitol; Drug: Gemcitabine (GEM) and Nab-paclitaxel

INTERVENTIONS:
Drug: Paricalcitol — Paricalcitol 12mcg, administered orally on every day of each 28-day cycle.
Drug: Gemcitabine (GEM) and Nab-paclitaxel — GEM (at 1,000 mg/m2) and Nab-paclitaxel (at 125 mg/m2 of bodysurface area), administered weekly for 3 of every 4 weeks (on days 1, 8 and 15 only).

SUMMARY:
The trial is designed to establish whether adding a vitamin D analogue, Paricalcitol, to standard chemotherapy treatment, Gemcitabine and Nab-paclitaxel, can improve the outcomes for patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This is an open-label phase II multi-centre single arm study which proposes to test the anti-tumour efficacy of paricalcitol, in combination with GEM/Nab-paclitaxel in patients with advanced metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedures.
2. Incurable recurrent, locally advanced or metastatic pancreatic adenocarcinoma.
3. Histologically or cytologically confirmed pancreatic adenocarcinoma.
4. No prior chemotherapy for incurable, locally advanced unresectable or metastatic pancreatic cancer. Patients may have received prior chemotherapy in the neo-adjuvant or adjuvant setting provided they have a minimum treatment-free interval of 3 months.
5. At least one measurable lesion according to RECIST criteria (Version 1.1). Patients with bone only disease are not eligible.
6. Aged 18 years or older
7. ECOG performance status 0 - 2
8. Adequate haematological, renal and hepatic function measured within 28 days prior to commencing study:

   * Total bilirubin ≤ ULN (or ≤ 3 x ULN (≤ grade 2) for patients with liver involvement)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (≤ grade

     1) (≤ 5 x ULN for patients with liver involvement by pancreatic cancer).
   * Glomerular filtration rate (GFR) ≥ 30mL/min/1.73 m2 (≤ grade 2) for patients with serum creatinine levels above or below the institutional normal range. If using creatinine clearance, actual body weight should be used for calculating creatinine clearance (e.g., using the Cockroft-Gault formula). For patients with a Body Mass Index (BMI) >30 kg/m2, lean body weight should be used instead.
   * Platelet count ≥ 100 x 109/L.
   * Haemoglobin (Hb) ≥ 8 g/dL (≤ grade 2)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (≤ grade 1)
   * Corrected serum calcium of ≤ 2.9 mmol/L (≤ grade 1).
9. Life expectancy of at least 12 weeks.
10. Women of childbearing potential and sexually active males must agree to use highly effective contraceptive measures. This applies from starting treatment until at least 6 months after the last study drug administration. The investigator or a designated associate is required to advise the patient how to achieve an adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

    i. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal). ii. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable). iii. Intrauterine device (IUD). iv. Intrauterine hormone-releasing system (IUS). v. Bilateral tubal occlusion. vi. Successfully vasectomised partner. vii. Sexual abstinence.

Exclusion Criteria:

1. Treated with other investigational drugs within 28 days or 5.5 half-lives of treatment start; in addition, concurrent alternative (complementary) medications are excluded within 28 days of treatment start.
2. Known brain metastases, unless previously treated and well-controlled for at least 2 months.
3. Dementia, altered mental status, or any other psychiatric condition that would interfere with the patient's safety or informed consent
4. History of other malignancy other than pancreatic cancer. However, patients who have been disease free from another malignancy for at least 5 years, or patients with a history of resected non-melanoma skin cancer or successfully treated in situ cancer and superficial bladder tumours (Ta, Tis, T1) are eligible.
5. Known history of hypercalcaemia.
6. Presence or history of symptomatic kidney stones in the last 5 years.
7. Active, clinically serious infections > grade 2 (CTCAE v5.0).
8. Greater than or equal to grade 2 sensory or motor neuropathy
9. Uncontrolled intercurrent illness, including, but not limited to uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or social situation that would affect compliance with the requirements of this study.
10. GI tract disease resulting in an inability to take oral medications, malabsorption syndrome, where previous surgical procedures affect absorption and uncontrolled inflammatory bowel disease.
11. History of diseases known to be associated with calcium disorders, including: ongoing hyperparathyroidism and Sarcoidosis.
12. Hypersensitivity to any of the excipients of gemcitabine, Nab-paclitaxel or Paricalcitol.
13. Known vitamin D toxicity
14. Undergoing treatment with the following therapies and medications:

    1. Concurrent use of drugs known to influence serum calcium such as thiazide diuretics, teriparatide (recombinant parathyroid hormone), calcitonin and multivitamin supplements containing > 400 IU of vitamin D or calcium.
    2. Current use of drugs which could influence bioavailability of paricalcitol (such as magnesium-containing antacids, bile-resin binders).
    3. Current use of strong inhibitors of CYP3A4 or CYP2C8.
    4. Current use of inducers of CYP3A4 or CYP2C8.
    5. Phosphate related medicinal products.

Note:

* Zoledronate or denosumab for patients with bone metastasis is allowed. Note patients with bone only disease are not eligible.
* Calcium intake is not restricted, but calcium supplementation is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 24 weeks from registration into the study
  PFS is the percentage of patients free of progression at 24 weeks from registration into the study as determined by radiographic disease assessments per RECIST version 1.1.
Overall survival (OS) | 18 months post last patient registered
  Overall survival (OS)

SECONDARY OUTCOMES:
Time to treatment failure | 18 months post last patient registered
  Time to Treatment Failure (TTF) is defined as time from registration to discontinuation of therapy or add-on of new anti-cancer therapy for any reason (including death, progression and toxicity).
Tumour response rate Duration of response | 18 months post last patient registered
  Confirmed tumour response rate as assessed by RECIST criteria version 1.1. Duration of response (DR) as assessed by RECIST criteria version 1.1.

OTHER OUTCOMES:
Safety and tolerability | 18 months post last patient registered
  Incidence of adverse events reported and toxicity evaluation as per the NCI CTCAE version 5.0
Incidence of hypercalcaemia | 18 months post last patient registered
  Incidence of hypercalcaemia

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Bryan Hennessy, Principal Investigator — Beaumont Hospital
Locations (6):
- Ireland (6):
  - Tallaght University Hospital, Dublin, Dublin 24
  - St. Vincent's University Hospital, Dublin, Dublin 4
  - Beaumont Hospital, Dublin, Dublin 9
  - Cork University Hospital, Cork
  - University Hospital Limerick, Limerick
  - University Hospital Waterford, Waterford